CLINICAL TRIAL: NCT05930860
Title: Efficacy and Safety of Endoscopic Submucosal Dissection for the Treatment of Superficial Gastric Neoplasms - An Italian Society of Digestive Endoscopy (SIED) Study
Brief Title: Efficacy and Safety of ESD for the Treatment of Superficial Gastric Neoplasms
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 4349
Record Dates: First submitted 2023-03-02; First posted 2023-07-05 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Gastric Cancer
Keywords: Endoscopic Submucosal Dissection; Endoscopic Resection
MeSH Terms: conditions — Stomach Neoplasms | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endoscopic Submucosal Dissection — Endoscopic Submucosal Dissection

SUMMARY:
Endoscopic submucosal dissection (ESD) is the technique that has replaced surgery in the treatment of early neoplastic lesions of the stomach (LNPS). ESD of LNPS allows: a) less invasiveness compared to surgery; b) greater chances of "en bloc" resection and R0 resection compared to mucosectomy for lesions larger than 15 mm. Recent 2015 ESGE guidelines provide precise recommendations for the use of ESD in the treatment of LNPS, but Italy lacks prospective data on the efficacy and safety of ESD in a large sample of patients. A multicenter prospective observational study to create a database on the use of ESD in LNPS is essential to provide information regarding the efficacy and safety of ESD in Italy. This database would also provide information regarding the criteria applied in the use of ESD in the treatment of early gastric neoplasia

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Endoscopic and histologic diagnosis of gastric superficial neoplasm that can be treated by ESD according to ESGE guidelines.
* Gastric neoplasm outside of latest ESD guidelines criteria in patients unfit for surgery

Exclusion Criteria:

* Final diagnosis of non neoplastic lesion.
* Gastric neoplasm outside of latest ESD guidelines criteria in patients fit for surgery
* Evidence of muscolar layer invasion or limph nodes or other organs metastasis at EUS or TC when performed.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients with gastric superficial neoplasms that can be treated by ESD according to ESGE guidelines or with gastric neoplasm outside of latest ESD guidelines criteria that are unfit for surgery.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-12-12 (Actual); Primary Completion 2025-08-12 (Estimated); Study Completion 2031-12-12 (Estimated)

PRIMARY OUTCOMES:
En bloc resection rate | 10 years
  removal of the lesion into a single piece.
R0 resection rate | 10 years
  complete removal of the tumor with histologically lateral and vertical margins of the specimen free from dysplasia
Curative resection rate | 10 years
  R0 resection with combined microstaging parameters not suggestive for high metastatic potential risk.
Complication rate | 10 years
  bleeding, perforation and stenosis.
Recurrence rate | 10 years
  dysplastic tissue at the site of resection at follow-up endoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Federico Barbaro, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Digestive Endoscopy Unit, Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Italy